CLINICAL TRIAL: NCT05487560
Title: A Multi-center, Prospective Cohort, Observational Study to Evaluate the Incidence of Major Adverse Cardiocerebrovascular Events According to Time Interval of Taking Medication in Patients With Acute Coronary Syndrome or Cerebral Infarction Who Received Dual AntiPlatelet Therapy (DAPT) for the Secondary Prevention and Esomezol Cap for the Prevention of Gastrointestinal Bleeding
Brief Title: An Observational Study to Evaluate the Incidence of MACCE According to Time Interval of Taking Medication in Patients With Acute Coronary Syndrome or Cerebral Infarction Who Received DAPT for the Secondary Prevention and Esomezol Cap for the Prevention of Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: HM-ESO-OS-01
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Acute Coronary Syndrome or B Cerebral Infarction Requiring DAPT(Clopidogrel + Aspirin) for at Least 6 Months
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 12-hour interval group (No interventional): DAPT(Clopidogrel + Aspirin) and Esomezol Cap taken every 12 hours
  Interventions: Drug: Esomezol Cap
- co-administration group (No interventional): Taking DAPT(Clopidogrel + Aspirin) and Esomezol Cap at the same time
  Interventions: Drug: Esomezol Cap

INTERVENTIONS:
Drug: Esomezol Cap — Esomezol Cap, Once daily administered per the locally approved product information

SUMMARY:
This study is to evaluate the incidence rate of Major Adverse CardioCerebrovascular Events(MACCE) in Patients with Acute Coronary Syndrome or Cerebral Infarction Who Received DAPT for the secondary prevention and Esomezol Cap for the prevention of gastrointestinal bleeding.

DETAILED DESCRIPTION:
This study was a multi-center, prospective, non-interventional, observational study of administering Esomezol Cap for the purpose of preventing gastrointestinal bleeding.

Data was collected from patients receiving routine treatment at hospitals in South Korea. Each patient visited the institution according to the protocol that designed the follow-up visits for six months to examine the safety of Esomezol Cap.

This study approved by the institutions' IRBs and was conducted in compliance with clinical research ethics regulations.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥19
2. Among patients who visited the hospital due to the onset or recurrence of acute coronary syndrome or cerebral infarction within 1 month prior to registration, patients who are expected to receive DAPT(Clopidogrel + Aspirin) for at least 6 months, in combination with Esomezol Cap for the purpose of preventing gastrointestinal bleeding Patients receiving or planning to receive treatment
3. Subject who can written informed consent voluntarily

Exclusion Criteria:

1) Patients for whom use of Esomezol Cap is prohibited

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Coronary Syndrome or B Cerebral Infarction requiring DAPT (Clopidogrel + Aspirin) for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 4133 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
The incidence of total Major Adverse CardioCerebrovascular Events(MACCE) from baseline | 6 months

SECONDARY OUTCOMES:
The incidence of MACCE by each of the following constituent variables | 6 months
  MACCE: Death due to cardiovascular abnormalities, myocardial infarction, stroke (ischemic or hemorrhagic), Target vessel reperfusion (in case of repeated intervention or coronary artery bypass surgery), All other cardiovascular events requiring hospitalization
The incidence e of Major bleeding | 6 months
  Major bleeding: intracranial hemorrhage, bleeding requiring a transfusion or A decrease in hemoglobin level ≥ 5 g/dL or a decrease in hematocrit ≥ 15%
The incidence of Minor bleeding | 6 months
  Minor bleeding: Any bleeding other than major bleeding
The incidence of GI Bleeding | 6 months
  GI Bleeding: hematemesis, melena/hematochezia, Fecal Occult Blood Test, FOBT
Occurrence and aspect of adverse events(AEs) | 6 months
Medication compliance evaluation | 6 months
Drug administration dose of DAPT(Clopidogrel + Aspirin) and Esomezol Cap | baseline
Drugs that are prescribed in combination other than DAPT(Clopidogrel + Aspirin) and Esomezol Cap for the treatment of patients with acute coronary syndrome or cerebral infarction | baseline
Add-on drugs for the treatment of patients with acute coronary syndrome or cerebral infarction | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi Pharmaceutical Company Limited, Seoul, South Korea